CLINICAL TRIAL: NCT03624907
Title: Consecutive Vs. Non-Consecutive Stereotactic Body Radiotherapy For Early Stage Non-Small Cell Lung Cancer
Brief Title: Daily vs. Non-Daily SBRT for NSCLC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Florida (Other)
Collaborators: DiaCarta, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201801625; OCR17400 (Other: University of Florida)
Record Dates: First submitted 2018-08-06; First posted 2018-08-10 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: stereotactic body radiotherapy (SBRT)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either daily or non-daily stereotactic body radiotherapy (SBRT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consecutive Daily Treatment (Other): Participant will receive daily stereotactic body radiotherapy at a dose of 48-50 Gy in 4-5 fractions with treatment occurring over 4-5 days
  Interventions: Radiation: Daily Stereotactic Body Radiotherapy
- Non-Consecutive Daily Treatment (Other): Participant will receive non-daily stereotactic body radiotherapy at a dose of 48-50 Gy in 4-5 fractions with treatment occurring over 8-12 days
  Interventions: Radiation: Non-Daily Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Daily Stereotactic Body Radiotherapy — After randomization, participants will receive daily standard of care doses of radiotherapy at treating physicians discretion.
  Arms: Consecutive Daily Treatment
Radiation: Non-Daily Stereotactic Body Radiotherapy — After randomization, participants will receive non-daily standard of care doses of radiotherapy at treating physicians discretion.
  Arms: Non-Consecutive Daily Treatment

SUMMARY:
The purpose of this study is to determine if stereotactic body radiotherapy (SBRT) on non-consecutive days will increase the chances of curing non-small cell lung cancer when compared to daily treatment.

DETAILED DESCRIPTION:
The purpose of this study is to determine if treatment with stereotactic body radiotherapy (SBRT) on non-consecutive days will improve the chance of curing non-small cell lung cancer compared to treatment with SBRT on consecutive days. In either case, the dose of radiation is the same. Non-consecutive treatments will be at least 40 hours apart and no more than 100 hours apart. The total course of treatment will be 8-12 days. Consecutive treatments will be daily over 4-5 days within one calendar week. The total course of treatment will be 4-5 days.

The study team will assess if DNA from the tumor can be found in the blood to determine which patients respond quickest to radiotherapy. These results will not be made available to participants and will not change treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age (no upper age limit).
* A diagnosis of non-small cell lung cancer, T1-2 N0 M0 either with histologic confirmation or with documented interval growth of the index lesion on two interval computed tomography (CT) chest scans and an SUVmax of the lesion ≥ 3.0 on a pretreatment PET scan.
* Patient must be deemed medically inoperable or refuse surgery.
* Radiographic evaluation of the mediastinum and distant sites with a CT scan of the chest and PET scan.
* For T2b N0 patients, radiographic evaluation of the brain with magnetic resonance imaging (MRI) of the brain unless the patient has contraindications to an MRI scan (in which case a CT scan of the head is necessary).
* For central T1 N0 and all T2 N0 patients, pathologic sampling (either via endobronchial ultrasound-guided biopsy [EBUS] or mediastinoscopy) of mediastinal lymph nodes is required.
* ECOG Performance Status 0-2.
* For women of childbearing potential, negative pregnancy test within 2 weeks prior to SBRT treatment.
* Patients must be deemed able to comply with the treatment plan and follow-up schedule.
* Patients must provide specific informed consent prior to study entry.
* Women of childbearing potential and male participants who are sexually active must use adequate contraception during treatment and for 6 weeks following treatment.

Exclusion Criteria:

* Prior history of radiation therapy to the thorax that would likely increase the risk of serious complications from the radiotherapy delivered on this protocol.
* Prior history of lung cancer.
* Currently taking disease-modifying rheumatoid drugs (DMRDs).
* Severe, active co-morbidity, defined as follows:
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects. Note, however, that coagulation parameters are not required for entry into this protocol.
* Prior organ transplant.
* Systemic lupus.
* Psoriatic arthritis.
* Known to be HIV positive. HIV-positive patients are known to have worse clinical outcomes, especially for local, regional, and distant cancer control. This poorer prognosis is thought to be secondary to a compromised immune system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Two-year control measured by CT (computerized tomography) scan | Two years
  Control defined as Less than 20% increase in the largest dimension of treated tumor measurable by CT
Two year control measured by PET (positron emission tomography) scan | Two years
  Control defined as PET imaging with uptake of a similar intensity as the pretreatment staging PET

SECONDARY OUTCOMES:
Document acute and late toxicity related to treatment | 2 years
  This will be assessed using the most recent version of the Common Terminology Criteria for Adverse Events (CTCAE).
Document patient-reported quality of life before, during, and after treatment | 2 years
  This will be done using quality of life surveys
Evaluate circulating tumor DNA | 2 years
  This will be done by collecting blood prior to, during, and after treatment
Overall Survival | 2 years
  Tracked through patient follow up
Progression Free Survival | 2 years
  Tracked through patient follow up

CONTACTS AND LOCATIONS:
Overall Officials: Anamaria Yeung, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Department of Radiation Oncology Davis Cancer Pavilion, Gainesville, Florida
  - University of Florida Health Proton Therapy Institute, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No